CLINICAL TRIAL: NCT05459272
Title: A Randomized, Placebo-Controlled Clinical Trial on a Dietary Supplement Containing Melatonin and Herbal Products to Improve Sleep Quality in Subjects With Insomnia Problems
Brief Title: Clinical Trial on a Food Supplement With Melatonin and Herbal Products to Improve Sleep Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uriach Consumer Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: URI-AQ-SUEFORT-2021
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-05

CONDITIONS: Sleep Disorders
Keywords: Sleep disorder,; Dietary supplement; Insomnia; Actigraphy
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This is a single-center, randomized, double-blind, placebo-controlled clinical trial with a dietary supplement with melatonin and herbal products, with two parallel group of subjects.
  Once the informed consent is signed, the patient will be assigned a patient code. The study treatment will be provided in white boxes with trial and patient identification labels, which will be identical for both products (dietary supplement and placebo), and the administration regimen will be the same for both products, thereby maintaining the double blind.
  Treatment intake will begin on study day 7 and end on day 14.
  The investigator will have an encrypted randomization list, so that, if necessary, he/she can determine the treatment group assigned to a patient.
  Treatment compliance will be recorded by the investigator at the 14-day visit.
  No other pharmacological or non-pharmacological treatment for insomnia will be allowed during the study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Aquilea Sueño Forte (Experimental): Patients included in this group will be administered dietary supplement with melatonin and herbal products, one tablet daily 30 min before to go to bed during 7 days (from day 7 to day 14).
  Interventions: Dietary Supplement: Aquilea Sueno Forte
- Control (Placebo Comparator): The control will consist of a placebo based on excipients without active ingredients so that the tablet has the same appearance as the test product.
  Patients should take one tablet daily 30 min before to go to bed during 7 days (from day 7 to day 14).
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Aquilea Sueno Forte — The test product consists of a dietary supplement in the form of tablets with three layers containing: melatonin (1.95 mg/tablet) and herbal products (extracts from Griffonia, Passiflora, California poppy, Valerian, Melissa).
  Patients should take one tablet daily 30 min before go to bed during 7 days (from day 7 to day 14).
  Arms: Experimental: Aquilea Sueño Forte
Other: Placebo — The placebo will consist of tablets with three layers and with the same appearance as the dietary supplement under study, but containing no active ingredients.
  Patients should take one tablet daily 30 min before go to bed during 7 days (from day 7 to day 14).
  Other Names: Control
  Arms: Control

SUMMARY:
A randomized, double-blind, placebo-controlled clinical trial on the ability of a dietary supplement containing melatonin and herbal products to improve sleep quality in subjects with insomnia problems with a 15-day follow-up period.

DETAILED DESCRIPTION:
This is a single-centre clinical trial on a dietary supplement with a 15-day follow-up period.

The investigators will include patients of legal age with DSM-5 diagnostic criteria for insomnia, without other sleep disorders.

The study will begin at baseline visit (day 0), when the inclusion and exclusion criteria will be confirmed and patient will sign the informed consent form. Information related to sleeping disorder will be collected and actigraphy device will be delivered to the patient. Patient will wear the device during 14 days.

After 7 days of wearing the device, patient will return to the follow-up visit (visit 1). The actigraph data will be downloaded and the treatment will be dispensed to the patient. Regimen will consist of taking one tablet per day of the product (dietary supplement or placebo) 30 minutes before bedtime during the following 7 days and will continue to wear the device.

At day 15 (final visit) patient will return the actigraph and clinical and safety data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients of legal age with DSM-5(*) diagnostic criteria for insomnia assessed from the Sleep Test responses (ST: 5-item questionnaire modified from the "Oviedo Sleep Questionnaire").
* Patients with insomnia of the following types: sleep onset insomnia (> 30 minutes of sleep latency), maintenance insomnia (frequent awakenings or inability to fall asleep after awakening) or mixed insomnia
* Patients who are not on treatment or have not taken any dietary supplements or hypnotics for insomnia, or any other psychoactive drug in the past week.
* Patients able to understand the implications of the study and who demonstrate this by voluntarily signing the informed consent

DSM-5 diagnostic criterion for insomnia:

A. A predominant complaint of dissatisfaction with sleep quantity or quality, associated with one (or more) of the following symptoms:

1. Difficulty initiating sleep. (In children, this may manifest as difficulty initiating sleep without caregiver intervention.)
2. Difficulty maintaining sleep, characterized by frequent awakenings or problems returning to sleep after awakenings. (In children, this may manifest as difficulty returning to sleep without caregiver intervention.)
3. Early-morning awakening with inability to return to sleep. B. The sleep disturbance causes clinically significant distress or impairment in social, occupational, educational, academic, behavioral, or other important areas of functioning.

C. The sleep difficulty occurs at least 3 nights per week. D. The sleep difficulty is present for at least 3 months. E. The sleep difficulty occurs despite adequate opportunity for sleep. F. The insomnia is not better explained by and does not occur exclusively during the course of another sleep-wake disorder (e.g., narcolepsy, a breathing-related sleep disorder, a circadian rhythm sleep-wake disorder, a parasomnia).

G. The insomnia is not attributable to the physiological effects of a substance (e.g., a drug of abuse, a medication).

H. Coexisting mental disorders and medical conditions do not adequately explain the predominant complaint of insomnia.

Exclusion Criteria:

* Pregnant or nursing women
* Patients with other sleep disorders: narcolepsy, obstructive apnea, circadian rhythm disorder, parasomnias
* Patients with active psychiatric disorders or cognitive impairment
* Patients with serious diseases that, in the physician's opinion, could interfere with the results of the study or disadvise their participation in it
* Patients who do not give their written consent
* Patients with known hypersensitivity or intolerance to any of the active ingredients or components of the dietary supplement or placebo.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-10 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in mean sleep latency (SL) | At the end of study (Day 15)
  Change in sleep latency comparing mean sleep latency during first week (without treatment) with mean sleep latency during second week (with treatment), assessed by actigraphy.
Change in total sleep time (TST) | At the end of study (Day 15)
  Change in total sleep time comparing mean total sleep time during first week (without treatment) with mean total sleep time during second week (with treatment), assessed by actigraphy.
Change in number of awakenings at night, assessed by actigraphy | At the end of study (Day 15)
  Change in number of awakenings at night comparing average number of awakenings at night during first week (without treatment) with average number of awakenings at night during second week (with treatment), assessed by actigraphy.
Change in distribution of sleep and awake periods throughout the day (DSW) | At the end of study (Day 15)
  Changes in distribution of sleep and awake periods throughout the day (DSW) comparing the DSW during first week (without treatment) with DSW during second week (with treatment), assessed by actigraphy.

SECONDARY OUTCOMES:
Type of insomnia | At the beginning
  Proportion of patients with each type of insomnia: conciliation insomnia, maintenance insomnia or mixed insomnia
Time from insomnia onset | At the beginning (Day 0)
  Time from insomnia problems onset (weeks, months)
Symptoms secundary to insomnia | At the beginning (Day 0)
  Mean of number of symptoms caused by insomnia: fatigue o discomfort, day time sleepiness, lack of memory or concentration, low performance, lack of energy, headache, gastrointestinal symptoms, irritability, concern about sleep.
Lack of memory or concentration secundary to insomnia | At the beginning (Day 0)
  Percentage of patients with lack of memory or concentration caused by insomnia.
Fatigue o discomfort secundary to insomnia | At the beginning (Day 0)
  Percentage of patients with fatigue o discomfort caused by insomnia.
Day time sleepiness secundary to insomnia | At the beginning (Day 0)
  Percentage of patients with day time sleepiness caused by insomnia.
Low performance secundary to insomnia | At the beginning (Day 0)
  Percentage of patients with low performance caused by insomnia.
Lack of energy secundary to insomnia | At the beginning (Day 0)
  Percentage of patients with lack of energy caused by insomnia.
Headache secundary to insomnia | At the beginning (Day 0)
  Percentage of patients with headache caused by insomnia.
Gastrointestinal symptoms secundary to insomnia | At the beginning (Day 0)
  Percentage of patients with gastrointestinal symptoms caused by insomnia.
Irritability secundary to insomnia | At the beginning (Day 0)
  Percentage of patients with irritability caused by insomnia.
Concern about sleep secundary to insomnia | At the beginning (Day 0)
  Percentage of patients with concern about sleep caused by insomnia.
Change in Pittsburgh Sleep Quality Index (PSQI) score | At the end of study (Day 15)
  Change in PSQI score comparing score obtained at the beginning (day 0) and at the end of the study (day 15)
Change in Insomnia Severity Index (ISI) score | At the end of study (Day 15)
  Change in Insomnia Severity Index (ISI) score comparing score obtained at the beginning (day 0) and at the end of the study (day 15)
Change in quality of life score (SF-12) | At the end of study (Day 15)
  Change in quality of life score (SF-12) comparing score obtained at the beginning (day 0) and at the end of the study (day 15)
Change in mean sleep latency (SL) according to electronic sleep diary | At the end of study (Day 15)
  Change in mean of SL (time it takes to fall asleep when you go to bed) comparing mean SL during first week (without treatment) with mean SL during second week (with treatment), according to electronic sleep diary
Change in number of awakenings at night, according to electronic sleep diary | At the end of study (Day 15)
  Change in number of awakenings at night comparing mean SL during first week (without treatment) with mean SL during second week (with treatment), according to electronic sleep diary
Change in total minutes awake out of bed, according to electronic sleep diary | At the end of study (Day 15)
  Change in mean of total minutes awake out of bed comparing mean of total minutes during first week (without treatment) with mean of total minutes during second week (with treatment), according to electronic sleep diary
Change in total minutes awake intrasleep, according to electronic sleep diary | At the end of study (Day 15)
  Change in mean of total minutes awake intrasleep comparing mean of total minutes during first week (without treatment) with mean of total minutes during second week (with treatment), according to electronic sleep diary
Tolerability and safety of the product | At the end of study (Day 15)
  Number of participants with incidence of treatment-related adverse effects and adverse reaction as a Measure of Safety and Tolerability
Compliance | At the end of study (Day 15)
  Number of days taking the treatment before going to sleep
Patient satisfaction | At the end of study (Day 15)
  Patient satisfaction on the efficacy and tolerability of treatment with the dietary supplement, using 5-point Likert scales ((0=very dissatisfied, 1=dissatisfied, 2=indifferent, 3=satisfied, 4=very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Escribá, PhD, Principal Investigator — Principal Investigator
Locations (1):
- Instituto de Medicina del Sueño, Alboraya, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No